CLINICAL TRIAL: NCT06211985
Title: Copeptın as a Dısease Severıty Indıcator: A Prospectıve Case-Control Study
Brief Title: Copeptin: Disease Severity Indicator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berker Okay (Other)
Responsible Party: Sponsor-Investigator, Berker Okay, M.D., Haseki Training and Research Hospital
Organization: Haseki Training and Research Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 63-2023
Record Dates: First submitted 2023-12-23; First posted 2024-01-18 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Lower Respiratory Tract and Lung Infections; Ventilator Lung; Bronchopneumonia; Bronchitis
MeSH Terms: conditions — Bronchopneumonia; Bronchitis

STUDY DESIGN:
Intervention Model Description: Blood tests were taken from all children included in the study to study the biomarker called 'Copeptin'.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bronchiolitis Group (Active Comparator): patients admitted to the ward with a diagnosis of Bronchiolitis (Group 1)
  Interventions: Diagnostic Test: Copeptin level measurement
- Mild to Moderate Pneumonia Group (Active Comparator): patients admitted to the ward with a diagnosis of mild to moderate pneumonia (Group 2)
  Interventions: Diagnostic Test: Copeptin level measurement
- Severe Pneumonia Group (Active Comparator): patients admitted to the ward with a diagnosis of severe pneumonia (Group 2)
  Interventions: Diagnostic Test: Copeptin level measurement
- Control Group (Active Comparator): the control group without pneumonia (Group 4)
  Interventions: Diagnostic Test: Copeptin level measurement

INTERVENTIONS:
Diagnostic Test: Copeptin level measurement — Throughout the study period, a total of 202 eligible patients were admitted to the hospital. Twenty-four patients were excluded due to lack of consent from their families, and an additional 103 patients were excluded based on the predefined exclusion criteria. In the control group, 72 individuals without chronic or acute diseases were initially eligible, but 46 of them were excluded due to lack of consent from their families. The study included patients who met the inclusion criteria and whose families provided consent, and it concluded upon reaching a total of 25 patients for each group. Additional blood samples were collected from each child within every group to assess copeptin levels, in conjunction with routine tests

SUMMARY:
Copeptin serves as a biomarker emanating from the pituitary gland, functioning as the precursor to arginine vasopressin (AVP). Its role in the regulation of endothelial dysfunction, inflammation, and water-electrolyte balance has been established. The measurement of AVP levels poses challenges due to its brief half-life and the intricate nature of its detection method. In contrast, copeptin provides an indirect means of gauging circulating AVP levels, as it can be conveniently assessed through a sandwich immunoassay. As a neuroendocrine stress hormone, copeptin emerges as a prognostic indicator, reflective of an individual's stress burden. Moreover, its applicability extends to various acute conditions such as ischemic stroke or myocardial infarction. Notably, copeptin proves to be a dependable tool in the differential diagnosis of diverse ailments characterized by polyuria and polydipsia.

Lower respiratory tract infection (LRTI) stands as the predominant cause of morbidity and mortality among children and adolescents globally. Notably, copeptin has demonstrated utility in forecasting the severity and complications associated with severe pneumonia in adults. While early investigations into copeptin's role in pediatric LRTI suggest its potential for diagnosing pneumonia and predicting complications, the outcomes of these studies present conflicting results.

Although there has been a notable increase in studies on copeptin in pediatric patients over the past decade, research specifically exploring its correlation with pneumonia remains scarce. This prospective case-control study is designed to investigate the potential association between copeptin levels and the severity of illness in pediatric patients with pneumonia. The study aims to determine whether copeptin levels can serve as a reliable predictor of disease severity in pneumonia, offering valuable insights for clinical application. The outcomes of this research may contribute significantly to our comprehension of copeptin's role in disease prognosis and management, thereby facilitating the development of more efficacious diagnostic and therapeutic approaches. Additionally, the study seeks to identify the factors influencing copeptin levels and establish a cut-off value for copeptin in pediatric patients diagnosed with pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with pneumonia,
* The family must have given informed consent for the study.

Exclusion Criteria:

* Individuals with underlying lung conditions (such as cystic fibrosis, bronchopulmonary dysplasia, asthma, bronchiectasis, tuberculosis),
* Individuals with underlying chronic illnesses (inclusive of heart, kidney, liver, gastrointestinal, and endocrine disorders),
* Individuals with obesity or malnutrition,
* Individuals with hyponatremia detected in their tests,
* Individuals with signs of dehydration,
* Individuals with a history of hospitalization within the last 72 hours.

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Predict disease severity in children with pneumonia with copeptin | 1 months
  Copeptin may hold promise as a predictor of disease severity in children with lower respiratory tract infections. It may show potential to guide physicians in determining the need for hospitalization and ventilator support.
  To measure this, patients were divided into groups and copeptin values of patients who needed ventilator support or who were hospitalized were compared with copeptin values of others using SPSS statistical program.

SECONDARY OUTCOMES:
Copeptin is more powerful than other acute phase reactants in predicting disease severity. | 1 months
  Copeptinin may perform better than other acute phase reactants such as neutrophil to lymphocyte ratio, fibrinogen to albumin ratio, c-reactive protein and procalcitonin in indicating the severity of the disease.
  To measure this, patients were divided into groups and copeptin values of patients who needed ventilator support or who were hospitalized were compared with copeptin values of others using SPSS statistical program.

CONTACTS AND LOCATIONS:
Locations (1):
- UHS Haseki Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Du JM, Sang G, Jiang CM, He XJ, Han Y. Relationship between plasma copeptin levels and complications of community-acquired pneumonia in preschool children. Peptides. 2013 Jul;45:61-5. doi: 10.1016/j.peptides.2013.04.015. Epub 2013 May 6. PMID 23659862
- [Background] Mohamed GB, Saed MA, Abdelhakeem AA, Salah K, Saed AM. Predictive value of copeptin as a severity marker of community-acquired pneumonia. Electron Physician. 2017 Jul 25;9(7):4880-4885. doi: 10.19082/4880. eCollection 2017 Jul. PMID 28894549
- [Background] Abdel-Fattah M, Meligy B, El-Sayed R, El-Naga YA. Serum Copeptin Level as a Predictor of Outcome in Pneumonia. Indian Pediatr. 2015 Sep;52(9):807-8. doi: 10.1007/s13312-015-0723-x. PMID 26519722
- [Background] Alcoba G, Manzano S, Lacroix L, Galetto-Lacour A, Gervaix A. Proadrenomedullin and copeptin in pediatric pneumonia: a prospective diagnostic accuracy study. BMC Infect Dis. 2015 Aug 19;15:347. doi: 10.1186/s12879-015-1095-5. PMID 26286191
- [Background] Wrotek A, Jackowska T, Pawlik K. Sodium and copeptin levels in children with community acquired pneumonia. Adv Exp Med Biol. 2015;835:31-6. doi: 10.1007/5584_2014_41. PMID 25252899
- [Background] Baumann P, Fuchs A, Gotta V, Ritz N, Baer G, Bonhoeffer JM, Buettcher M, Heininger U, Szinnai G, Bonhoeffer J; ProPAED study group. The kinetic profiles of copeptin and mid regional proadrenomedullin (MR-proADM) in pediatric lower respiratory tract infections. PLoS One. 2022 Mar 10;17(3):e0264305. doi: 10.1371/journal.pone.0264305. eCollection 2022. PMID 35271609